CLINICAL TRIAL: NCT00149201
Title: Randomized Phase III Study of 5-FU Continuous Infusion (5FUci) Versus MTX+5-FU Sequential Therapy (MF) in Gastric Cancer With Peritoneal Metastasis (JCOG0106-MF, MF/5FU)
Brief Title: A Study of 5-FU Versus MTX+5-FU in Gastric Cancer With Peritoneal Metastasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Japan Clinical Oncology Group, Japan Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0106-MF; C000000123
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Cancer; Neoplasm Metastasis
Keywords: gastric cancer; peritoneal metastasis; randomized trial; 5-FU; MTX
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 5-FU continuous infusion
Drug: MTX + 5-FU sequential therapy

SUMMARY:
To develop effective chemotherapy regimen against gastric cancer with peritoneal metastasis

DETAILED DESCRIPTION:
Peritoneal metastasis is common in advanced gastric cancer and is considered an incurable disease state. Peritoneal metastasis may cause serious complications, such as intestinal obstruction, massive ascites, and hydronephrosis associated with the clinical presentation of abdominal pain and fullness, vomiting, constipation, malnutrition and renal dysfunction.5-FU continuous infusion remains the mainstay for chemotherapy against gastric cancer. On the other, sequential MTX+5-FU was reported to be effective in advanced gastric cancer with peritoneal metastasis in some phase II studies. Therefore, the randomized phase III study of 5-FU versus sequential MTX+5-FU in gastric cancer with peritoneal metastasis was conducted.

ELIGIBILITY:
Inclusion Criteria:

1. histologic confirmation of gastric adenocarcinoma
2. inoperable metastatic disease or recurrent metastatic disease after surgery
3. disease with peritoneal metastasis
4. 20 years or more but less than 75 years
5. performance status 2 or less on the Eastern Cooperative Oncology Group scale
6. no prior treatment for gastric carcinoma except for surgery and adjuvant chemotherapy
7. no prior chemotherapy or radiotherapy for other disease except for gastric cancer
8. adequate bone marrow function, adequate liver function, and adequate renal function
9. no prior transfusion for anemia
10. provision of written informed consent

Exclusion Criteria:

1. Massive pleural effusion
2. brain metastasis with symptoms
3. severe diarrhea
4. other severe medical conditions (infection, diabetes, hypertension, acute myocardial infarction, unstable angina, liver cirrhosis, intestinal pneumonia, pulmonary fibrosis)
5. other active malignancies

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
oral intake
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Kuniaki Shirao, MD,PhD, Study Chair — Gatrointestinal Oncology Division, National Cancer Center Hospital
Locations (34):
- Japan (34):
  - Aichi Cancer Center Hospital, 1-1,Kanokoden,Chikusa-ku,Nagoya, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, 18,Kuriyado,Kake-machi,Okazaki, Aichi-ken
  - Nagoya Medical Center, 4-1-1,Sannomaru,Naka-ku,Nagoya, Aichi-ken
  - Aomori Prefectural Central Hospital, 2-1-1,Higashitsukurimiti,Aomori, Aomori
  - National Cancer Center Hospital East, 6-5-1,Kashiwanoha,Kashiwa, Chiba
  - Chiba Cancer Center Hospital, 666-2,Nitona-cho,Chuo-ku,Chiba, Chiba
  - Asahi General Hospital, I-1326,Asahi, Chiba
  - National Hospital Organization Shikoku Cancer Center, 13,Horinouchi,Matsuyama, Ehime
  - Kyushu University Hospital, 3-1-1,Maidashi,Higashi-ku, Fukuoka
  - National Kyushu Cancer Center, 3-1-1,Notame,Minami-ku,Fukuoka, Fukuoka
  - Federation of national public service personnel mutual aid associations Tonan Hospital, Kita 1 Nishi 6,Chuo-ku,Sapporo, Hokkaido
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Hyogo Medical Center for Adults, 13-70,Kitaouji-cho,Akashi, Hyōgo
  - Kobe University Graduate School of Medicine, 7-5-2,Kusunoki-cho,Chuo-ku,Kobe, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, 6528,Koibuchi,Tomobemachi,Nishi-ibarakigun, Ibaraki
  - Iwate Prefectural Central Hospital, 1-4-1,Ueda,Morioka, Iwate
  - Kanagawa Cancer Center, 1-1-2,Nakao,Asahi-ku,Yokohama, Kanagawa
  - Kitasato University East Hospital, 2-1-1,Asamizodai,Sagamihara, Kanagawa
  - Yokohama City University Medical Center, 4-57,Urafunecho,Minami-ku,Yokohama, Kanagawa
  - Yokohama Mucipical Citizen's Hospital, 56,Okazawa-cho,Hodogaya-ku,Yokohama, Kanagawa
  - Kochi Health Science Center, 2125-1,Ike,Kochi, Kochi
  - Kumamoto Regional Medical Center Hospital, 5-16-10,Honjo,Kumamoto, Kumamoto
  - Kyoto University Hospital, 54,Syogoinkawara,Sakyo-ku,Kyoto, Kyoto
  - Tohoku University Hospital, 1-1,Seiryo-machi,Aoba-ku,Sendai, Miyagi
  - Saku Central Hospital, 197,Usuda,Saku, Nagano
  - Osaka Medical College, 2-7,Daigakucho,Takatsuki, Osaka
  - Saitama Medical School Hospital, 38,Morohongo,Moroyama-machi,Iruma-gun, Saitama
  - Saitama Cancer Center, 818,Komuro,Ina,Kita-adachi, Saitama
  - Sizuoka Cancer Center, 1007,Shimonagakubo,Nagaizumi-cho,Sunto-gun, Shizuoka
  - Tochigi Cancer Center, 4-9-13,Yohnan,Utsunomiya, Tochigi
  - Showa University School of Medicine, 1-5-8,Hatanodai,Shinagawa-ku, Tokyo
  - Cancer Institute Hospital, 3-10-6,Ariake,Koto-ku, Tokyo
  - National Cancer Center Hospital, 5-1-1 Tsukiji, Chuo-ku, Tokyo
  - Yamagata Prefectural Central Hospital, 1800,Aoyagi,Yamagata, Yamagata

REFERENCES:
- See also: Related Info — http://www.jcog.jp/